CLINICAL TRIAL: NCT06537713
Title: Diagnostic Role of Serum Testican and Ubiquitin Levels in Patients With Head Trauma
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramiz Yazıcı, Assistant Professor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019/159
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Moderate Traumatic Brain Injury; Testican-1; Ubiquitin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: The control group consisted of healthy individuals without any disease who voluntarily participated in the study.
  Interventions: Diagnostic Test: Testican-1
- Patients Group: The study specifically included patients over 18 years of age with moderate TBI (GCS: 9-13) who provided informed consent.
  Interventions: Diagnostic Test: Testican-1

INTERVENTIONS:
Diagnostic Test: Testican-1 — Testican-1 and ubiquitin can serve as early indicators for diagnosing worsening clinical course and mortality in patients with moderate traumatic brain injury.
  Other Names: Ubiquitin

SUMMARY:
We aimed to determine if testican-1 and ubiquitin can serve as early indicators for diagnosing worsening clinical course (presence of intraparenchymal pathology) and mortality in patients with moderate traumatic brain injury.

DETAILED DESCRIPTION:
The study specifically included patients over 18 years of age with moderate TBI (GCS: 9-13) who provided informed consent. The control group consisted of healthy individuals without any disease who voluntarily participated in the study. Patients with moderate TBI were divided into two groups: those with intracranial pathology (Subdural hemorrhage, epidural hemorrhage, subarachnoid hemorrhage, intraparenchymal hemorrhage, and contusion) and those without. Treatment was initiated according to ATLS in patients with moderate TBI, and blood samples taken at the time of admission to the emergency department were placed in Ethylenediaminetetraacetic acid (EDTA) tubes. The relationship between the patient's clinical scoring (GCS, ISS and AIS), brain CT results, and mortality status with testican-1 and ubiquitin levels was compared.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old
* having a GCS score between 9 and 13

Exclusion Criteria:

* under 18 years of age
* had missing data
* were pregnant
* had neurodegenerative disease
* had Central Nervous System (CNS) infection
* had cerebral palsy
* had penetrating head injury (by a cutting or piercing tool such as a firearm, knife, axe)
* patients with severe (GCS: 3-8) or mild (GCS: 14-15) TBI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with head trauma were categorized into three groups based on their GCS score: severe (3-8), moderate (9-13), and mild (14-15). The study specifically included patients over 18 years of age with moderate TBI (GCS: 9-13) who provided informed consent. Patients who were under 18 years of age, had missing data, were pregnant, had neurodegenerative disease, had Central Nervous System (CNS) infection, had cerebral palsy, or had penetrating head injury (by a cutting or piercing tool such as a firearm, knife, axe), as well as patients with severe (GCS: 3-8) or mild (GCS: 14-15) TBI, were not included in the study. The control group consisted of healthy individuals without any disease who voluntarily participated in the study. Patients with moderate TBI were divided into two groups: those with intracranial pathology (Subdural hemorrhage, epidural hemorrhage, subarachnoid hemorrhage, intraparenchymal hemorrhage, and contusion) and those without.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of testican-1 and ubiquitin levels in patients with moderate traumatic brain injuries and a control group | The study was conducted with blood samples taken at the time of admission.
  We compared the plasma blood levels of biomarkers in both groups

SECONDARY OUTCOMES:
ROC curve analysis for the prediction of intraparenchymal pathology (+) | The study was conducted with blood samples taken at the time of admission.
  We investigated the diagnostic value of biomarkers in detecting pathology on brain CT in patients with moderate traumatic brain injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni SUltan Suleyman Training and Research Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be shared upon reaching the corresponding author.

REFERENCES:
- [Background] Maas AIR, Menon DK, Manley GT, Abrams M, Akerlund C, Andelic N, Aries M, Bashford T, Bell MJ, Bodien YG, Brett BL, Buki A, Chesnut RM, Citerio G, Clark D, Clasby B, Cooper DJ, Czeiter E, Czosnyka M, Dams-O'Connor K, De Keyser V, Diaz-Arrastia R, Ercole A, van Essen TA, Falvey E, Ferguson AR, Figaji A, Fitzgerald M, Foreman B, Gantner D, Gao G, Giacino J, Gravesteijn B, Guiza F, Gupta D, Gurnell M, Haagsma JA, Hammond FM, Hawryluk G, Hutchinson P, van der Jagt M, Jain S, Jain S, Jiang JY, Kent H, Kolias A, Kompanje EJO, Lecky F, Lingsma HF, Maegele M, Majdan M, Markowitz A, McCrea M, Meyfroidt G, Mikolic A, Mondello S, Mukherjee P, Nelson D, Nelson LD, Newcombe V, Okonkwo D, Oresic M, Peul W, Pisica D, Polinder S, Ponsford J, Puybasset L, Raj R, Robba C, Roe C, Rosand J, Schueler P, Sharp DJ, Smielewski P, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Temkin N, Tenovuo O, Theadom A, Thomas I, Espin AT, Turgeon AF, Unterberg A, Van Praag D, van Veen E, Verheyden J, Vyvere TV, Wang KKW, Wiegers EJA, Williams WH, Wilson L, Wisniewski SR, Younsi A, Yue JK, Yuh EL, Zeiler FA, Zeldovich M, Zemek R; InTBIR Participants and Investigators. Traumatic brain injury: progress and challenges in prevention, clinical care, and research. Lancet Neurol. 2022 Nov;21(11):1004-1060. doi: 10.1016/S1474-4422(22)00309-X. Epub 2022 Sep 29. PMID 36183712
- [Background] Hossain I, Rostami E, Marklund N. The management of severe traumatic brain injury in the initial postinjury hours - current evidence and controversies. Curr Opin Crit Care. 2023 Dec 1;29(6):650-658. doi: 10.1097/MCC.0000000000001094. Epub 2023 Oct 11. PMID 37851061
- [Background] Shultz SR, Shah AD, Huang C, Dill LK, Schittenhelm RB, Morganti-Kossmann MC, Semple BD. Temporal proteomics of human cerebrospinal fluid after severe traumatic brain injury. J Neuroinflammation. 2022 Dec 8;19(1):291. doi: 10.1186/s12974-022-02654-0. PMID 36482407
- [Background] Hossain I, Marklund N, Czeiter E, Hutchinson P, Buki A. Blood biomarkers for traumatic brain injury: A narrative review of current evidence. Brain Spine. 2023 Dec 14;4:102735. doi: 10.1016/j.bas.2023.102735. eCollection 2024. PMID 38510630
- [Background] Silvestro S, Raffaele I, Quartarone A, Mazzon E. Innovative Insights into Traumatic Brain Injuries: Biomarkers and New Pharmacological Targets. Int J Mol Sci. 2024 Feb 17;25(4):2372. doi: 10.3390/ijms25042372. PMID 38397046
- [Background] Kim DS, Kim GW. Biofluid-based Biomarkers in Traumatic Brain Injury: A Narrative Review. Brain Neurorehabil. 2024 Mar 18;17(1):e8. doi: 10.12786/bn.2024.17.e8. eCollection 2024 Mar. PMID 38585027
- [Background] Iseki K, Hagino S, Zhang Y, Mori T, Sato N, Yokoya S, Hozumi Y, Goto K, Tase C. Altered expression pattern of testican-1 mRNA after brain injury. Biomed Res. 2011 Dec;32(6):373-8. doi: 10.2220/biomedres.32.373. PMID 22199127
- [Background] Yakovlev AG, Faden AI. Mechanisms of neural cell death: implications for development of neuroprotective treatment strategies. NeuroRx. 2004 Jan;1(1):5-16. doi: 10.1602/neurorx.1.1.5. PMID 15717003
- [Background] Tongaonkar P, Chen L, Lambertson D, Ko B, Madura K. Evidence for an interaction between ubiquitin-conjugating enzymes and the 26S proteasome. Mol Cell Biol. 2000 Jul;20(13):4691-8. doi: 10.1128/MCB.20.13.4691-4698.2000. PMID 10848595
- [Background] Azar S, Hasan A, Younes R, Najdi F, Baki L, Ghazale H, Kobeissy FH, Zibara K, Mondello S. Biofluid Proteomics and Biomarkers in Traumatic Brain Injury. Methods Mol Biol. 2017;1598:45-63. doi: 10.1007/978-1-4939-6952-4_3. PMID 28508357
- [Background] Liu MC, Akinyi L, Scharf D, Mo J, Larner SF, Muller U, Oli MW, Zheng W, Kobeissy F, Papa L, Lu XC, Dave JR, Tortella FC, Hayes RL, Wang KK. Ubiquitin C-terminal hydrolase-L1 as a biomarker for ischemic and traumatic brain injury in rats. Eur J Neurosci. 2010 Feb;31(4):722-32. doi: 10.1111/j.1460-9568.2010.07097.x. PMID 20384815
- [Background] Welch RD, Ayaz SI, Lewis LM, Unden J, Chen JY, Mika VH, Saville B, Tyndall JA, Nash M, Buki A, Barzo P, Hack D, Tortella FC, Schmid K, Hayes RL, Vossough A, Sweriduk ST, Bazarian JJ. Ability of Serum Glial Fibrillary Acidic Protein, Ubiquitin C-Terminal Hydrolase-L1, and S100B To Differentiate Normal and Abnormal Head Computed Tomography Findings in Patients with Suspected Mild or Moderate Traumatic Brain Injury. J Neurotrauma. 2016 Jan 15;33(2):203-14. doi: 10.1089/neu.2015.4149. Epub 2015 Dec 18. PMID 26467555
- [Background] Papa L, Lewis LM, Silvestri S, Falk JL, Giordano P, Brophy GM, Demery JA, Liu MC, Mo J, Akinyi L, Mondello S, Schmid K, Robertson CS, Tortella FC, Hayes RL, Wang KK. Serum levels of ubiquitin C-terminal hydrolase distinguish mild traumatic brain injury from trauma controls and are elevated in mild and moderate traumatic brain injury patients with intracranial lesions and neurosurgical intervention. J Trauma Acute Care Surg. 2012 May;72(5):1335-44. doi: 10.1097/TA.0b013e3182491e3d. PMID 22673263
- [Background] Mondello S, Kobeissy F, Vestri A, Hayes RL, Kochanek PM, Berger RP. Serum Concentrations of Ubiquitin C-Terminal Hydrolase-L1 and Glial Fibrillary Acidic Protein after Pediatric Traumatic Brain Injury. Sci Rep. 2016 Jun 20;6:28203. doi: 10.1038/srep28203. PMID 27319802